CLINICAL TRIAL: NCT00241683
Title: Fetal Growth Restriction & Maternal Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberta Ness, Dean, SPH, Dean - School of Public Health, The University of Texas Health Science Center, Houston
Other Study IDs: 1307; 5R01HL076532-03 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine whether or not women with a history of having a baby with intrauterine growth retardation (IUGR) was more likely to have risk factors for cardiovascular disease versus women with a pregnancy not complicated by IUGR.

DETAILED DESCRIPTION:
BACKGROUND:

Intrauterine growth restriction leads to major neonatal morbidity and mortality. Moreover, recent birth registry studies have suggested that women bearing IUGR babies may have an elevated risk of cardiovascular disease.

DESIGN NARRATIVE:

This cohort study tested whether exposed women, with a previous intrauterine growth restriction (IUGR) baby, versus unexposed women, with a pregnancy not complicated by IUGR, had elevations in markers of cardiovascular risk. Exposure was defined among a geographically defined cohort as having had a singleton baby in the < 5 %tile of weight for gestational age, in the absence of pre-pregnancy diabetes., hypertension, renal disease, or hypertension in pregnancy; controls had a singleton in the > 20%tile. Four to twelve years postpartum, women were assessed for multiple markers of cardiovascular risk, including blood pressure, lipids, adiposity, glucose and insulin, homocysteine and folate, markers of inflammation, markers of endothelial function, markers of angiogenesis, and markers of vascular function. Data analysis consisted of ANOVA and ANCOVA analyses comparing the outcomes of cardiovascular markers among exposed and unexposed women.

ELIGIBILITY:
Inclusion criteria:

* women 4 to 12 years after delivery of singleton infant
* women who gave birth between 1997 and 2002 at Magee-Womens Hospital in Pittsburgh, Pennsylvania

Exclusion criteria:

* women who had preeclampsia
* women who had prepregnancy hypertension
* women who had diabetes
* women who were currently pregnant or reported a prepregnancy chronic condition

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who were 4 to 12 years postpartum
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2005-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 to 12 years after pregnancy
Triglycerides and LDL cholesterol | 4 to 12 years after pregnancy

SECONDARY OUTCOMES:
Glucose | 4 to 12 years after pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Roberta B. Ness, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Result] Catov JM, Dodge R, Yamal JM, Roberts JM, Piller LB, Ness RB. Prior preterm or small-for-gestational-age birth related to maternal metabolic syndrome. Obstet Gynecol. 2011 Feb;117(2 Pt 1):225-232. doi: 10.1097/AOG.0b013e3182075626. PMID 21252733
- [Result] McClure CK, Bodnar LM, Ness R, Catov JM. Accuracy of maternal recall of gestational weight gain 4 to 12 years after delivery. Obesity (Silver Spring). 2011 May;19(5):1047-53. doi: 10.1038/oby.2010.300. Epub 2010 Dec 16. PMID 21164507
- [Result] McClure CK, Catov J, Ness R, Schwarz EB. Maternal visceral adiposity by consistency of lactation. Matern Child Health J. 2012 Feb;16(2):316-21. doi: 10.1007/s10995-011-0758-0. PMID 21404071